CLINICAL TRIAL: NCT01063049
Title: Gatorade/Miralax With or Without Bisacodyl vs NuLytely for Colonoscopy Preparation
Brief Title: Gatorade/Miralax With or Without Bisacodyl Versus NuLytely for Colonoscopy Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gastroenterology Services, Ltd. (Other)
Responsible Party: Principal Investigator, David Gerard, M.D., MD, Gastroenterology Services, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1220100180
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Preparation for Colonoscopy
MeSH Terms: interventions — gatorade; polyethylene glycol 3350; Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nulytely (Active Comparator): Nulytely (or Trilyte) 128 oz (1 gallon) to be consumed from about 5 PM to 9 PM the night before the colonoscopy.
  Interventions: Drug: NuLytely
- Gatorade/Miralax + Placebo (Experimental): Gatorade 64 oz (1/2 gallon), Miralax 306 g and a placebo (two 0.4 mg folic acid pills) to be consumed the day before the colonoscopy as follows: Miralax 51 g and placebo at 12 noon. Gatorade 64 oz mixed with Miralax 255 g from about 5 PM to 9 PM.
  Interventions: Drug: Gatorade/Miralax; Drug: Placebo
- Gatorade/Miralax + Bisacodyl (Experimental): Gatorade 64 oz (1/2 gallon), Miralax 306 g and Bisacodyl 10 mg (two 5 mg pills) to be consumed the day before the colonoscopy as follows: Miralax 51 g and Bisacodyl 10 mg at 12 noon. Gatorade 64 oz mixed with Miralax 255 g from about 5 PM to 9 PM.
  Interventions: Drug: Gatorade/Miralax; Drug: Bisacodyl

INTERVENTIONS:
Drug: Gatorade/Miralax — Gatorade 64 oz (1/2 gallon), Miralax 306 g to be consumed the day before your colonoscopy as follows: Miralax 51 g at 12 noon. Gatorade 64 oz mixed with Miralax 255 g from about 5 PM to 9 PM.
  Arms: Gatorade/Miralax + Bisacodyl; Gatorade/Miralax + Placebo
Drug: NuLytely — Nulytely (or Trilyte) 128 oz (1 gallon) to be consumed from about 5 PM to 9 PM the night before the colonoscopy.
  Arms: Nulytely
Drug: Bisacodyl — Bisacodyl 10 mg (two 5 mg pills) to be consumed the day before the colonoscopy at 12 noon.
  Arms: Gatorade/Miralax + Bisacodyl
Drug: Placebo — Placebo (two 0.4 mg folic acid pills) to be consumed the day before the colonoscopy
  Arms: Gatorade/Miralax + Placebo

SUMMARY:
The purpose of this study is to compare Nulytely (or Trilyte) with a Gatorade and Miralax combination for cleaning out the colon before colonoscopy. A laxative pill called Bisacodyl may also be used with the Gatorade and Miralax to see if it helps with the clean out process. We are trying to find out if either of these methods is more acceptable to the patient and does a better job cleaning out the colon for a colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old planning to undergo an elective colonoscopy.

Exclusion Criteria:

1. Patients who are allergic or intolerant to any on the study drugs.
2. Pregnant patients.
3. Patients who required multiple day colon preparation in the past.
4. Patients with ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or toxic megacolon would not be considered elective colonoscopies and are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Gerard, M.D., Principal Investigator — Gastroenterology Services, Ltd.
Locations (1):
- Gastroenterology Services, Downers Grove, Illinois, United States

REFERENCES:
- [Result] Gerard DP, Holden JL, Foster DB, Raiser MW. Randomized Trial of Gatorade/Polyethylene Glycol With or Without Bisacodyl and NuLYTELY for Colonoscopy Preparation. Clin Transl Gastroenterol. 2012 Jun 21;3(6):e16. doi: 10.1038/ctg.2012.11. PMID 23238266
- See also: On line publication of study resulting from this work. — http://www.nature.com/ctg/journal/v3/n6/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects had their colonoscopy performed between February 2010 and February 2011 by one of three gastroenterologists (DG, JH, and MR) with 17 to 34 years of experience. Colonoscopies were scheduled to begin between 0800 h and noon in the gastrointestinal labs at our office or two community hospitals.
Period: Overall Study
Arm/Group | Nulytely | Gatorade/Miralax + Placebo | Gatorade/Miralax + Bisacodyl
Started | 200 | 200 | 200
Completed | 200 | 200 | 200
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nulytely | Gatorade/Miralax + Placebo | Gatorade/Miralax + Bisacodyl | Total
Number analyzed (Participants) | 200 | 200 | 200 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 120 | 120 | 360
  >=65 years | 80 | 80 | 80 | 240
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (13.2) | 59.7 (13.8) | 61.3 (12.5) | 60.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 91 | 99 | 271
  Male | 119 | 109 | 101 | 329
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 200 | 600

OUTCOME MEASURES:

1. Primary Outcome: The Quality of the Colon Preparation Will be Graded Using the Boston Bowel Preparation Scale
Description: The Boston Bowel Preparation Scale measures cleanliness of the colon on a scale of 0 (very poor) to 9 (excellent).
Time Frame: After Colonoscopy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nulytely | Gatorade/Miralax + Placebo | Gatorade/Miralax + Bisacodyl
Number analyzed (Participants) | 200 | 200 | 200
units on a scale | 7.86 (1.55) | 8.05 (1.28) | 7.99 (1.41)

2. Secondary Outcome: The Ottawa Scale for Colonoscopy Preparation Will be Reported and Compared Among the 3 Groups to Allow for Comparisons to Some of the Older Literature
Description: Ottawa scale measures colon cleanliness on a scale from 14 (very poor) to 0 (excellent).
Time Frame: After Colonoscopy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nulytely | Gatorade/Miralax + Placebo | Gatorade/Miralax + Bisacodyl
Number analyzed (Participants) | 200 | 200 | 200
units on a scale | 2.80 (2.24) | 2.58 (2.47) | 2.71 (2.47)

ADVERSE EVENTS:
Time Frame: up to 1 month after colonoscopy.
Arm/Group | Nulytely | Gatorade/Miralax + Placebo | Gatorade/Miralax + Bisacodyl
Serious Adverse Events (participants affected / at risk) | 0/200 | 1/200 | 0/200
Other Adverse Events (participants affected / at risk) | 0/200 | 0/200 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nulytely (N=200) | Gatorade/Miralax + Placebo (N=200) | Gatorade/Miralax + Bisacodyl (N=200)
post-polypectomy bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Both the BBPS and OPS suffer from poorly designed scoring systems that are not easily converted into the poor/fair/good/excellent subjective rating scale, which is often used by gastroenterologists in their colonoscopy reports.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No